CLINICAL TRIAL: NCT05301556
Title: Effect of a Food for Special Medical Purpose (FSMP) Product During the Perioperative Period in Patients With Digestive Tract Tumor
Brief Title: Food for Special Medical Purpose in Patients With Digestive Tract Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BL43
Record Dates: First submitted 2022-02-15; First posted 2022-03-29 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Product (Experimental): Food for Special Medical Purpose (FSMP) is a special medical food for patients with tumors
  Interventions: Other: Experimental Product
- Control Product (Active Comparator): Nutrition Emulsion (TPF-T) TPF-T is a tumor-specific enteral nutrition therapy
  Interventions: Other: Control Product

INTERVENTIONS:
Other: Experimental Product — * Before the surgery: FSMP provides daily target energy needed by participants
  * 1-2 days after surgery: Start FSMP and advance as tolerated to achieve 20% of the daily target energy needed by participants
  * 3rd-5th day after surgery: Gradually increase FSMP intake every day as tolerated to provide 30-80% of the daily target energy needed by participants
  * 6th to 11th day after surgery. FSMP provides daily target energy needed by participants
  Arms: Experimental Product
Other: Control Product — * Before surgery: TPF-T provides daily target energy needed by participants
  * 1-2 days after surgery: Start TPF-T and advance as tolerated to achieve 20% of the daily target energy needed by participants
  * 3rd-5th day after surgery: Gradually increase TPF-T intake every day as tolerated to provide 30-80% of the daily target energy needed by participants
  * 6th to 11th day after surgery. TPF-T provides daily target energy needed by participants
  Arms: Control Product

SUMMARY:
This is a prospective, randomized, controlled, unblinded, parallel, multicenter, and non-inferiority study to demonstrate the safety and efficacy of a Food for Special Medical Purpose product (FSMP) in participants with digestive tract tumor undergoing surgical resection during the perioperative period.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, unblinded, parallel, and multicenter, and non-inferiority study to demonstrate the safety and efficacy of a FSMP in participants with digestive tract tumor undergoing surgical resection during the perioperative period. Half of the participants will receive FSMP, the other half will receive Enteral Nutrition Emulsion (TPF-T) as an active control.

Prealbumin, albumin, C-reactive protein (CRP), immunology parameters, vital signs, nutrition and safety-related laboratory parameters, compliance, and Adverse Events (AEs) will be evaluated in this study, to demonstrate its parity with TPF-T on efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Participant is male or female, between 18 and 75 years old, female participant is non-pregnant or non- lactating, at least 6 weeks postpartum
* Participants with digestive tract tumors diagnosed by histological method or radiological diagnosis and scheduled to undergo surgical resection
* Participant with NRS-2002 score ≥3
* Participant is willing to comply with the study protocol, able and willing to consume study product according to the protocol
* Participants with Body Mass Index 18.5 - 30 kg/m2
* Participant has voluntarily signed and dated an informed consent form (ICF), approved by an Institutional Review Board (IRB) / Independent Ethics Committee (IEC) prior to any participation in the study

Exclusion Criteria:

* Participant has an expected life expectancy < 3 months
* Participant has contraindications to enteral nutrition (such as active gastrointestinal hemorrhage, bowel obstruction, decompensated short bowel syndrome, high flow intestinal fistula, severe intraperitoneal infection, severe gastrointestinal emptying disorder, unstable vital signs, dyscoagulation, severe nausea, vomiting and/or uncontrolled diarrhea/steatorrhoea) that in the opinion of the study physician cannot be corrected
* Participant used parenteral nutrition or had plasma infused, RBC infused, albumin infused, amino acid infused or undergone radiotherapy and/or chemotherapy within 1 week before screening
* Participant with serum Albumin <2.5g/dl at the time of the screening
* Participant has moderate to severe anemia, i.e. Hgb < 90g / L
* Patients who plan to receive endoscopic tumor resection or / and palliative surgery
* Participant has renal dysfunction (serum creatinine > 2 times the upper limit of normal (ULN))
* Participant has liver insufficiency [serum alanine transaminase (ALT) and/or aspartate transaminase (AST) > 2 times the ULN or severe cholestasis (conjugated bilirubin > 2 times the ULN)]
* Participant has severe cardiac insufficiency (e.g., Severe arrhythmia or atrial fibrillation; myocardial ischemia or stent surgery with unstable cardiac function within 3 months prior to screening visit )
* Participant states that he/she has had a significant cardiovascular and cerebrovascular event (e.g., myocardial infarction, stroke) within six months prior to screening visit; or stated history of congestive heart failure
* Participant with type I diabetes, or type II diabetes with fasting blood glucose ≥8mmol/L
* Participant has history of significant neurological or psychiatric disorder
* Participant has history of alcoholism, drug abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures
* Participant has a known history of allergy or intolerance to any ingredient in the investigational products
* Participant is currently undergoing tumor immunotherapy taking medications/substances that could profoundly modulate appetite, metabolism or inflammatory level

  1. Appetite enhancers, pregnancy promoters, steroids (nasal inhalation, topical and optical steroids are acceptable);
  2. Anti-inflammatory fat emulsions or other oral nutritional supplementations/drugs containing Omega-3 fatty acids, protein, glutamine, or arginine.
  3. Dexamethasone, growth hormone or other drugs affecting metabolism;
* Participant is currently undergoing tumor immunotherapy or taking medications/substances that could profoundly modulate immune function, such as PD1 or PDL1 inhibitors; CTLA-4 inhibitor; Thymosin; Azathioprine; Cyclosporine; Tacrolimus; Tumor necrosis factor antagonist; Lentinan; immune-modulating Chinese medicine
* Participant with active tuberculosis and HIV infection
* Participant participated in any clinical trial within four weeks prior to the screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Serum Pre-Albumin | Baseline to Post Op Day (POD) 9
  Change in pre-albumin

SECONDARY OUTCOMES:
Serum Albumin | Baseline to Post Op Day (POD) 9
  Change in albumin
Weight | Baseline to Post Op Day (POD) 9
  Change in weight
Nutritional Risk Screening (NRS) 2002 | Baseline to Post Op Day (POD) 9
  NRS-2002 scored from 0 Low Risk to 7 High Risk

OTHER OUTCOMES:
C-reactive Protein (CRP) | Baseline to Post Op Day (POD) 9
  Change in CRP
Length of hospital stay | From Date of Admission until Date of Discharge, typically up to 14 days
  Days stay in hospital
Hand Grip Strength | Baseline to Post Op Day (POD) 9
  Measured in kg
Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline to Post Op Day (POD) 9
  Healthcare Professional assessed score with range from 0 to 5; higher scores indicate worsening functional status
Product Intake | Baseline to Post Op Day (POD) 9
  Daily volume of study product consumed
Adverse Events | Baseline to Post Op Day (POD) 9
  Reported adverse events for assessment of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Shengqi Li, PhD, Study Chair — Abbott Nutrition
Locations (8):
- China (8):
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - The Six Afffilated Hospital Sun Yat-sen University, Guangzhou
  - The Affiliated Hospital of Qingdao University, Qingdao

IPD SHARING:
Plan to Share IPD: No